CLINICAL TRIAL: NCT05173090
Title: Influence of Intra-abdominal Ropivacaine 0.5% Spray on Postoperative Analgesia in Laparoscopic Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, MD, Principal investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ropicoelio
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Appendectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaïne 0,5% (Active Comparator): 3 mg/kg of ropivacaine 0.5% sprayed into the abdominal cavity
  Interventions: Drug: Ropivacaïne 0,5% for appendectomy or cholecystectomy surgery
- NaCl 0,9% (Placebo Comparator): NaCl 0,9% sprayed into the abdominal cavity
  Interventions: Drug: Ropivacaïne 0,5% for appendectomy or cholecystectomy surgery

INTERVENTIONS:
Drug: Ropivacaïne 0,5% for appendectomy or cholecystectomy surgery — Visual analog scale 15 min after arrival in the recovery room, then H+4, H+6, H+12, H+24 and one week after the operation

SUMMARY:
Assessing postoperative pain after ropivacin 0.5% spray in the abdominal cavity during laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Appendectomy or cholecystectomy surgery

Exclusion Criteria:

* Allergy to local anesthetics
* Intolerance to tramadol HCl
* Patient with peritonitis
* Pregnant women
* Surgery without laparoscopy
* Chronic pain before the operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Patient's pain | During appendectomy and cholecystectomy surgery
  The patient's satisfaction was assessed by visual analog scale, ranging from one (worse outcome )to four (better outcome